CLINICAL TRIAL: NCT02837211
Title: The TREND Study: Tapered Reduction in Energy Intake as a Novel Approach to Dieting
Acronym: TREND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00037795
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tapered Diet (Experimental)
  Interventions: Behavioral: Tapered Low Calorie Diet
- Traditional Low Calorie Diet (Active Comparator)
  Interventions: Behavioral: Traditional Low-Calorie Diet

INTERVENTIONS:
Behavioral: Tapered Low Calorie Diet — All participants will start with a 3 week run-in period during which they are fed a diet at 1.4 x their resting metabolic rate (kcal). Participants who are weight stable at the end of run in and are randomized to the Tapered Diet Arm will undergo the following 24 week feeding study intervention.
  The difference between a participant's run-in period energy intake and low-calorie "prescribed" energy intake (1000 kcal for women; 1200kcal for men) will be divided by six. At weekly intervals from weeks 1-6, daily caloric intake will be decreased by this fixed amount, reaching the final daily caloric goal (1000 kcals for women and 1200 kcals for men) by the end of the 6th week. Participants will present twice per week during weeks 1-6 to receive food that sums to that week's prescribed calorie level.
  From weeks 7-24, these participants will then follow a traditional low-calorie diet, still presenting for food pickups twice per week at a stable caloric level during this period.
  Arms: Tapered Diet
Behavioral: Traditional Low-Calorie Diet — All participants will start with a 3 week run-in period during which they are fed a diet at 1.4 x their resting metabolic rate (kcal). Participants who are weight stable at the end of run in and are randomized to the Traditional Diet Arm will undergo the following 24 week feeding study intervention.
  Immediately following run-in, these participants will start a low-calorie diet (1000 kcal per day for women; 1200kcal for men) Participants will present twice per week during weeks 1-24 to receive food that sums to that week's prescribed calorie level.
  Arms: Traditional Low Calorie Diet

SUMMARY:
TREND is a pilot randomized trial comparing two alternative methods of initiating a low-calorie weight loss diet. The study will compare the traditional diet initiation of abruptly dropping energy intake to 1000 kcal/day for women and 1200 kcal/day for men versus a 6 week tapering of energy intake from a baseline level. These two approaches will be compared with respect to their impact on energy regulatory systems of the body, weight loss and other measures, up to a year after diet initiation.

DETAILED DESCRIPTION:
Diets are the mainstay of many obesity treatment programs, yet they fail for a variety of reasons. Patients find it difficult to comply with caloric restriction during active weight loss, and to adhere to long-term changes that promote weight loss maintenance. Underlying these difficulties are a number of physiologic changes enacted by the body in response to energy restriction. These changes promote increased hunger, decreased satiety and slowed metabolic rate, making diet compliance and sustained weight loss very difficult. From the body's perspective, a rapid and substantial drop in caloric intake may represent a metabolic emergency, and it responds accordingly, in an attempt to maintain body weight.

Weight loss results only from achieving and maintaining a large energy deficit, but it is not known whether the initiation phase of diets would be more likely to promote success if it were done gradually, in the form of a caloric taper. We hypothesize that, by slowly introducing a prescribed caloric restriction over a period of 1-2 months (rather than using an immediate drop in calories), the body's homeostatic response to energy restriction might be blunted or circumvented, resulting in lower levels of hunger, improved satiety, and better preservation of metabolic rate during diet initiation - all factors that would promote adherence and successful weight loss.

To test this hypothesis, the investigators will conduct a pilot randomized feeding trial comparing two types of low-calorie diets with similar macronutrient composition. Although both diets will ultimately rely on similar caloric deficits to produce weight loss, they will differ at the point of diet initiation. The following will be compared: (1) a traditional diet, where the entire energy deficit is initiated immediately; and (2) a "caloric taper" diet, during which participants will be gradually reduced from baseline levels of energy consumption to the lower calorie level required for weight loss, over a 6-week period.

After a 2-week run-in to establish equilibrium weight among 40 eligible persons, 30 obese adults will be randomized to the 2 study arms and follow them for 52 weeks. We will compare the two groups with respect to the following outcomes, measured in terms of change from baseline (week 0) levels:

1. Circulating levels of the orexogenic hormone, Ghrelin, at weeks 1, 6, 12, 24, and 52;
2. Circulating levels of the "satiety" hormones, Leptin and Glucagon-like Peptide (GLP-1) at weeks 1, 6, 12, 24, and 52;
3. Body composition, as assessed with dual energy x-ray absorptiometry, at 24 and 52 weeks;
4. Resting metabolic rate as assessed by indirect calorimetry at 24 and 52 weeks;
5. Change in body weight (kg) and body mass index (kg/m2) at weeks 6,12, 24 and 52;
6. Self-reported hunger (using VAS) and compliance with program at weeks 1, 6, 12, 24 and 52.
7. Change in weight-related quality of life, using the IWQOL-LITE at weeks 12, 24, and 52.

Hypothesis: patients in the "taper" arm will experience less activation of body regulatory systems designed to oppose weight loss, with similar weight loss by 24 weeks and greater weight loss maintenance by 52 weeks, compared to "traditional low-calorie diet" arm patients.

ELIGIBILITY:
Inclusion Criteria:

* Employee of Wake Forest Baptist Medical Center
* BMI 30-40 kg/m2
* Interested in weight loss
* <90 min/wk of exercise at baseline
* Receives medical care through Wake Forest and has WakeOne account

Exclusion Criteria:

* Already participating in another diet or weight loss program or research study
* History of bariatric surgery
* History of eating disorder
* History of cancer (other than non-melanomatous skin cancer)
* History of thyroid disease
* History of severe mental illness
* Diagnosis of diabetes
* Currently pregnant, breastfeeding or planning pregnancy
* Peri or post-menopausal
* Food allergies or sensitivities
* Vegetarian
* Night Shift worker
* Planning prolonged travel in next 6-8 months or frequent out of town travel
* on any medication that could promote weight loss or weight gain

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Ghrelin | change from baseline at weeks 1, 6, 12, 24, 52
  Orexogenic hormone
Leptin | change from baseline at weeks 1, 6, 12, 24, 52
  Satiety hormone

SECONDARY OUTCOMES:
Glucagon-like peptide-1 (GLP1) | change from baseline at weeks 1, 6, 12, 24, 52
  Satiety hormone
Body Composition (percent body fat, percent lean mass) | change from baseline at week 24 and 52
  Assessed with DEXA Scan
Resting Metabolic Rate (RMR) | change from baseline at weeks 12, 24, 52
  Assessed with indirect calorimetry
Weight (kg) | Change from baseline at weeks 6, 12, 24 and 52
Hunger | weeks 1, 6, 12, 24, 52
  Visual-analogue scale, self report
Weight-related quality of life (IWQOL-Lite) | Change from baseline at weeks 12, 24, and 52
  Validated survey measure

CONTACTS AND LOCATIONS:
Overall Officials: Kristina H Lewis, MD MPH SM, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States